CLINICAL TRIAL: NCT02665845
Title: Combination Corticosteroids+5-aminosalicylic Acids Compared to Corticosteroids Alone in the Treatment of Moderate-severe Active Ulcerative Colitis: A Protocol of a Multi-center Prospective Randomized Investigator Blinded Trial.
Brief Title: Combination Corticosteroids+5-aminosalicylic Acids Compared to Corticosteroids Alone (for Ulcerative Colitis).
Acronym: COMBOMESA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1508090; 2015-002671-21 (EudraCT Number)
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-ASA group (Experimental): Patients will receive corticosteroids with optimized 5-ASA.
  Interventions: Drug: 5-ASA; Drug: Corticosteroids
- Control group (Active Comparator): Patients will receive corticosteroids alone.
  Interventions: Drug: Corticosteroids

INTERVENTIONS:
Drug: 5-ASA — 5ASA treatment (oral 5ASA will be given to all patients in this arm, in addition to topical 5ASA in patients who tolerate it).
  Other Names: 5-aminosalicylates
  Arms: 5-ASA group
Drug: Corticosteroids — Corticosteroids will be given to all patients.
  Other Names: Usual care

SUMMARY:
The role of steroids in the treatment of severe ulcerative colitis (UC) exacerbation is well established and recommended by professional societies. Similarly, 5-aminosalycilates (5-ASA) agents in the form of mesalamine/mesalzine are well established proven therapy in mild-moderate UC, and the combination of oral 5-ASA with topical (per-rectal enema) 5-ASA was shown to be superior to oral 5ASA alone in patients with mild moderate UC. Thus, in most cases, when a patient with UC experiences a flare while taking 5-ASA therapy, treatment is usually optimized by maximizing the oral dose to 4gr/day and adding topical therapy until the flare is controlled. If this is unhelpful, or if the flare is severe to begin with, corticosteroids are usually prescribed. However, there are very scarce data comparing steroids versus 5-ASA in the treatment of severe UC exacerbation.

The aim of this study is to compare the efficacy of steroids alone vs. combination of steroids + 5-ASA in the treatment of moderate-severe UC exacerbation.

DETAILED DESCRIPTION:
The role of steroids in the treatment of severe ulcerative colitis (UC) exacerbation is well established and recommended by professional societies. This recommendation is based on pivotal studies carried 50-60 years ago, by Truelove &Witts. Similarly, 5-aminosalycilates (5-ASA) agents in the form of mesalamine/mesalzine are well established proven therapy in mild-moderate UC, and the combination of oral 5-ASA with topical (per-rectal enema) 5-ASA was shown to be superior to oral 5ASA alone in patients with mild moderate UC. Thus, in most cases, when a patient with UC experiences a flare while taking 5-ASA therapy, treatment is usually optimized by maximizing the oral dose to 4gr/day and adding topical therapy until the flare is controlled. If this is unhelpful, or if the flare is severe to begin with, corticosteroids are usually prescribed. However, there are very scarce data comparing steroids versus 5-ASA in the treatment of severe UC exacerbation. In 1962 truelove et al compared topical and systemic corticosteroid therapy with sulphasalazine, and found steroids to be superior to sulfasalazine. Importantly, there are no data investigating whether the addition and/or continuation of 5-ASA agents as combination therapy with systemic corticosteroids is superior to corticosteroids alone in patients with moderate-severe active UC. This knowledge gap is pronounced in patients admitted to the hospital for intravenous corticosteroid treatment with moderate severe UC flare, in whom it is currently unknown if the addition of 5-ASA (Oral and/or topical) to corticosteroids will confer additional benefit and improve patients outcomes. Thus, in practical terms, the decision whether to stop or continue 5-ASA treatment or whether to add 5-ASA to steroids in the treatment of moderate-severe UC exacerbation is taken on an arbitrary basis. This is important shortcoming and knowledge gap in current medicine, as patients admitted with moderate-severe UC flare who do not respond to corticosteroids and require salvage therapy with infliximab, cyclosporine, or even urgent colectomy. This makes it prudent to explore any avenue for possible improvement of response to corticosteroids in this setting, for instance by addition of 5ASA.

The aim of this study is: To compare the efficacy of steroids alone vs. combination of steroids + 5-ASA in the treatment of moderate- severe UC exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* UC known and diagnosed by established clinical-endoscopic and histological criteria or newly-diagnosed UC, based on clinical and endoscopic findings, and about to start treatment with corticosteroids.
* Current hospitalization with Severe UC exacerbation as defined by a Lichtiger score of >10
* Age >18
* Has not been on oral systemic corticosteroids more than 14 days prior to hospitalization
* If taking a thiopurine, the dose need to be stable for the last 2 months before admission

Exclusion Criteria:

* Pregnant women
* Allergy / unable to take prednisone / hydrocortisone/ 5-ASA.
* Active infection - either enteric or elsewhere
* Severe renal, liver or cardio respiratory comorbidity
* Toxic megacolon, or clinical features suggestive of a need for imminent colectomy
* Treatment with an anti-TNF within the prior 3 months
* Prior treatment with cyclosporine or tacrolimus within the prior 3 months
* Alcohol dependency
* Unable or unwilling to provide informed consent
* Participating in other clinical trial within the 2 months prior to admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who respond to the treatment by day 7. | Day 7
  The primary endpoint will be the percentage of patients who respond to the treatment by day 7. Response will be defined by a drop of >3 points in the lichtiger score and an absolute score <10 on the two prior consecutive days without the need for rescue medications or surgery. In patients who improve and are discharged prior to day 7, the lichtiger score will be calculated based on the two last days of hospitalization, provided that at least 3 days of study medications were dispensed. Patients discharged before 3 days of study medications have been administered will be considered in-eligible and will be dropped out of the analyses.

CONTACTS AND LOCATIONS:
Overall Officials: ROBLIN Xavier, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (6):
- Chu Saint Etienne, Saint-Etienne, France
- Department of Gastroenterology Venizeleio General Hospital, Leoforos Knosou, Heraklion, Greece
- Sheba Medical Center, Tel Litwinsky, Ramat-Gan, Israel
- Università di Roma Sapienza, Rome, Italy
- Zvezdara University Clinical Center, Gastroenterology Department, Belgrade, Serbia
- Institute of Gastroenterology and Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No